CLINICAL TRIAL: NCT00356603
Title: Imigran STATdose - Japan Clinical Experience Study for Self-injection
Brief Title: Study Of Sumatriptan Succinate Injection Kit In Patients With Migraine or Cluster Headache In Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STA106711
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Migraine Disorders
Keywords: Migraine; Sumatriptan Succinate Injection Kit; Cluster Headache; self-injection
MeSH Terms: conditions — Migraine Disorders; Cluster Headache | interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sumatriptan (Experimental): Sumatriptan
  Interventions: Drug: Sumatriptan Succinate

INTERVENTIONS:
Drug: Sumatriptan Succinate — Sumatriptan Succinate

SUMMARY:
This study will be conducted to collect cases treated by self-injection of sumatriptan 3mg kit product for the treatment of migraine or cluster headache attacks in clinical settings, to demonstrate the efficacy, and to examine patient acceptability (simplicity and usefulness) and rate of successful self-injection.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of migraine (with or without aura) or cluster headache according to the International Classification of Headache Disorders, Version 2 (ICHD-II)
* History of migraine or cluster headache persisting for at least 6 months
* Migraine: One to 6 attacks of moderate or severer headaches per month during the 2 months prior to enrollment
* Cluster Headache: Each attack persisting for at least 45 minutes
* Written informed consent obtained from the patient. When a patient is a minor, written informed consent from his/her proxy consenter (e.g., person with parental authority) will also be required.

Exclusion criteria:

* History of hypersensitivity to any of the ingredients of 5-HT1B/1D receptor antagonists (e.g., triptans) or serious AE due to treatment with these drugs
* History of serious adverse event attributable to treatment with Imigran® Injection 3
* History of myocardial infarction, current or previous history of ischemic heart disease or its symptoms/signs, or current history of atypical variant angina (coronary arteriospasm)
* Previous history of cerebrovascular disorder or transient cerebral ischemic attack
* Current or previous history of peripheral angiopathy (including Raynaud's syndrome)
* Systolic blood pressure (SBP) >160 mmHg or diastolic blood pressure (DBP) >95 mmHg at the start of treatment period
* Current familial hemiplegic migraine, basilar migraine, or sporadic hemiplegic migraine
* Current abuse of ergotamine- or dihydroergotamine-containing preparations or triptans
* Pregnant women, lactating mothers, women who may be pregnant, or women of childbearing potential using no appropriate contraceptive measures.
* Epilepsy or organic cerebral disorder which may lead to convulsion
* Previous history of hypersensitivity to sulfonamides
* Known drug allergy or idiosyncrasies
* Known drug dependency or alcoholism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-06-20 (Actual); Primary Completion 2006-08-07 (Actual); Study Completion 2006-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Japan (4):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 20 June 2006 to 07 August 2006 across four centers in Japan.
Pre-assignment Details: A total of 75 participants with history of migraine or cluster headache persisting for at least 6 months had entered into the study.
Groups:
- Migraine: Participants with migraine administered one subcutaneous dose of Sumatriptan Succinate Injection 3 milligrams (mg) kit product (0.5 milliliter [mL] containing 4.2 mg of sumatriptan succinate) by self-injection. The recommended injection site was the thigh.
- Cluster Headache: Participants with cluster headache administered one subcutaneous dose of Sumatriptan Succinate Injection 3 mg kit product (0.5 mL containing 4.2 mg of sumatriptan succinate) by self-injection. The recommended injection site was the thigh.
Period: Overall Study
Arm/Group | Migraine | Cluster Headache
Started | 39 | 36
Completed | 33 | 33
Not Completed | 6 | 3
Not completed — Other | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Migraine: Participants with migraine administered one subcutaneous dose of Sumatriptan Succinate Injection 3 mg kit product (0.5 mL containing 4.2 mg of sumatriptan succinate) by self-injection. The recommended injection site was the thigh.
- Total: Total of all reporting groups
Arm/Group | Migraine | Cluster Headache | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.2 (9.9) | 37.4 (9.0) | 39.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 8 | 34
  Male | 7 | 25 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 33 | 33 | 66
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Headache Relief at 60 Minutes Post Dose(Migraine) or 30 Minutes Post Dose(Cluster Headache)
Description: Headache relief rate was the percentage of participants who showed effectiveness 60 minutes post dose (migraine) or 30 minutes post dose (cluster headache). Data for participants with percentage effectiveness along with 95% confidence interval has been presented.
Time Frame: 30 minutes or 60 Minutes after each administration
Population: Full Analysis Set (FAS) Population included patients who self-administered the study product and have at least one efficacy data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Migraine + Cluster Headache: Participants with migraine and cluster headache administered one subcutaneous dose of Sumatriptan Succinate Injection 3 mg kit product (0.5 mL containing 4.2 mg of sumatriptan succinate) by self-injection. The recommended injection site was the thigh.
Arm/Group | Migraine | Cluster Headache | Migraine + Cluster Headache
Number analyzed (Participants) | 33 | 33 | 66
Percentage of participants | 93.9 [79.8 to 99.3] | 93.9 [79.8 to 99.3] | 93.9 [85.2 to 98.3]

2. Secondary Outcome: Number of Participants With Subject-rated Acceptability of the Sumatriptan 3mg Kit Product
Description: The subject-rated acceptability of sumatriptan succinate injection 3 mg kit product had three questions, question 1 was "Was the kit product easy to use?", question 2 was "Do you want to use the kit product in the future?" and question 3 was "Do you consider that the kit product is necessary for the treatment of your illness?". The responses were given as yes or no. Data for number of participants who responded to the three questions as yes or no has been presented.
Time Frame: Up to 2 months
Population: FAS Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Migraine | Cluster Headache | Migraine + Cluster Headache
Number analyzed (Participants) | 33 | 33 | 66
Participants
  Question 1: Yes | 32 | 33 | 65
  Question 1: No | 1 | 0 | 1
  Question 2: Yes | 31 | 31 | 62
  Question 2: No | 2 | 2 | 4
  Question 3: Yes | 31 | 29 | 60
  Question 3: No | 2 | 4 | 6

3. Secondary Outcome: Percentage of Participants With Investigator/Sub Investigator-rated Successful Self-injection Rate
Description: The investigator/sub investigator-rated successful self-injection rate was the percentage of participants who were able to use the kit as directed by the investigator/ sub investigator. The response was given as yes or no. Data for percentage of participants who were actually able to use the kit as directed has been presented.
Time Frame: Up to 2 months
Population: FAS Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Migraine | Cluster Headache | Migraine + Cluster Headache
Number analyzed (Participants) | 33 | 33 | 66
Percentage of participants | 100 | 100 | 100

ADVERSE EVENTS:
Time Frame: All Adverse events and serious adverse events that occurred after administration of the investigational product (including the day of administration) and before last participant last visit were analyzed (approximately 2 months).
Description: Safety Population was used for the analysis of safety data. Safety population consisted of patients who received at least one dose of study medication.
Arm/Group | Migraine | Cluster Headache | Migraine + Cluster Headache
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/66
Other Adverse Events (participants affected / at risk) | 5/33 | 10/33 | 15/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Migraine (N=33) | Cluster Headache (N=33) | Migraine + Cluster Headache (N=66)
Malaise (General disorders) | 1 | 2 | 3
Nausea (Gastrointestinal disorders) | 1 | 2 | 3
Blood creatine phosphokinase increased (Investigations) | 0 | 3 | 3
Asthenia (General disorders) | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2
Somnolence (Nervous system disorders) | 1 | 1 | 2
Chest discomfort (General disorders) | 0 | 2 | 2
Feeling abnormal (General disorders) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
White blood cell count increased (Investigations) | 0 | 1 | 1
Protein urine present (Investigations) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.